CLINICAL TRIAL: NCT03780114
Title: Knowledge, Attitude and Practice Survey for Group of Egyptian Dentists About Infection Control in Different Pediatric Dental Clinics: A Cross-Sectional Study
Brief Title: Knowledge, Attitude and Practice Survey for Egyptian Dentists About Infection Control in Pediatric Dental Clinics
Acronym: case-only
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noha Hany Hassan Khalil Hassan, Principal investigator, Cairo University
Other Study IDs: CEBD-CU-2018-11-17
Record Dates: First submitted 2018-12-07; First posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Infection Control

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- interns: intern pediatric dentists

SUMMARY:
This study is designed to gather information about knowledge of pediatric dentistry interns towards infection control procedures in pediatric dental clinics, also about their attitude towards the rules and guidelines of infection control, and finally their practice to these guidelines to achieve the ultimate infection control in pediatric dental clinics.

DETAILED DESCRIPTION:
Patient's safety is considered a very important medical protocol which aims at improving quality of patient's care, minimizing treatment mistakes and improving safety to the maximum extent that can be reached. On this approach infection is one of the most critical issues in healthcare service worldwide, where it can be transmitted during dental procedures through direct and indirect contact , in addition to high risk blood borne infections , and nowadays we are facing global emergence and re-emergence of many communicable diseases that can also be transmitted during dental practice.

As a result of the high risk of transmission of the above infections, high standard precautions must be implemented for all patients attending dental clinics regardless of their infection status , because those patients could be in the prodromal phase or carriers without even knowing. In addition, some infectious diseases have prolonged incubation periods during which antibodies can't be detected , So in order to avoid infection transmission hazards and to achieve patient's safety, infection prevention and control of cross-contamination are our goal in providing a secure environment for patients and healthcare workers within healthcare settings in general and more specifically in dental practices.

Transmission of infectious agents among patients and dental health care personnel (DHCP) in dental settings is rare. However, transmissions in dental settings, including patient-to-patient transmissions, have been documented. In most cases, investigators failed to link a specific lapse of infection prevention and control with a particular transmission. However, reported breakdowns in basic infection prevention procedures included unsafe injection practices, failure to heat sterilize dental handpieces between patients, and failure to monitor autoclaves by conducting spore tests.

Generally, Concerns have increased considerably by a report about the transmission of human immunodeficiency virus (HIV) from an American dentist to five of his patients. With the presence of people infected with hepatitis B and C and the HIV viruses, cross infection has become a major concern for dentists, dental personnel and patients. On the other hand, developing countries including Egypt showed the increased prevalence of transmission of infection among dental clinics.

Therefore, Universal precautions should be followed considering all patients as infectious. However, Most hospitals have no infection control programs due to the lack of awareness of the problem or absence of properly trained personnel. This highlight the need for training to improve understanding of principles, practices, and implementation, in addition to the conditions that cause disease transmission, So all dental settings, regardless of the level of care provided, must make infection prevention a priority and should be equipped to observe Standard Precautions and other infection prevention recommendations contained in CDC's Guidelines for Infection Control in Dental Health-Care Settings - 2003.

POS format:

P (population): Interns in pediatric dental clinics.

O (outcome): Knowledge, attitude, and practice of infection control in pediatric dental clinics.

* Outcome measuring tool: A Questionnaire.
* Outcome measuring unit: Closed- ended questions (dichotomous, multiple choice questions, Likert, and matrix questions).

S (study design): Cross-sectional survey (Observational type of study).

Research question:

What is the level of knowledge, attitude, and practice of intern pediatric dentists in pediatric dental clinics in Faculty of Dentistry, Cairo University towards infection control protocols and guidelines in pediatric dentistry?

ELIGIBILITY:
Inclusion Criteria:

* Interns working in pediatric dental clinics who have ended their rounds in faculty of Dentistry, Cairo University

Exclusion Criteria:

* interns and dentists who refuse to participate in the study.
* interns who are not performing regular attendance in the pediatric dental clinics.

Ages: 23 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: • Interns who have ended their pediatric dentistry rounds will be asked to answer the questionnaire.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-02-01 (Estimated); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
Knowledge | 1 month
  closed- ended questionnaire , 16 knowledge questions, if the total number of participants answered all the questions this will be mentioned, and if any was not answered or missed for any reason this will be reported.

OTHER OUTCOMES:
Attitude | 1 month
  closed- ended questionnaire, 8 questions, if the total number of participants answered all the questions this will be mentioned, and if any was not answered or missed for any reason this will be reported.
Practice | 1 month
  closed- ended questionnaire, 36 questions, if the total number of participants answered all the questions this will be mentioned, and if any was not answered or missed for any reason this will be reported.

IPD SHARING:
Plan to Share IPD: Undecided